CLINICAL TRIAL: NCT00792233
Title: Improved Understanding of the Biology and Use of TNF Inhibition in Children With JIA
Brief Title: Determining Predictors of Safe Discontinuation of Anti-TNF Treatment in JIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P60 AR047784-Project 2; P60AR047784 (NIH)
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Poly JIA; TNF; Remission
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants taking anti-TNF medications will be monitored for signs of their disease for 6 months. If, after 6 months, their disease has become inactive, they will stop taking anti-TNF medications for up to 8 months. If participants who are no longer taking anti-TNF medications have a disease flare-up, they will begin treatment again.
  Interventions: Other: Withdrawal of anti-TNF therapy

INTERVENTIONS:
Other: Withdrawal of anti-TNF therapy — Anti-TNF therapy will be discontinued at the third visit in children who demonstrate persistent inactive disease for at least 6 months.

SUMMARY:
Polyarticular juvenile idiopathic arthritis (Poly JIA) is a form of juvenile arthritis, which is a chronic disease affecting approximately 250,000 people younger than 16 years of age. Poly JIA can be treated with anti-tumor necrosis factor (anti-TNF), a type of medication that is often effective but also has some toxic side effects and is expensive. Among those with poly JIA who are effectively treated with anti-TNF, some can remain healthy off the medication, but some begin to feel the effects of their disease again once the medication is stopped. This study will attempt to find whether certain tests or signs can predict which people with poly JIA can safely stop their anti-TNF medications.

DETAILED DESCRIPTION:
Juvenile arthritis is a chronic disease affecting approximately 250,000 people younger than 16 years of age in the United States. Its symptoms include swelling, pain, and damage in the joints. Juvenile arthritis can take four different forms, including poly JIA. Poly JIA affects five or more joints, generally the smaller ones in wrists and fingers, causing stiffness, joint damage, and sometimes eye inflammation in the children and adolescents who suffer from it. Approximately 30% of people with juvenile arthritis have Poly JIA.

Treatment for juvenile arthritis involves drugs with escalating strength, depending on what each individual responds to best. The first treatment option is non-steroidal anti-inflammatory drugs (NSAIDs), such as Motrin IB and Aleve. The second treatment option is methotrexate (MTX). About 30% to 50% of poly JIA patients are effectively treated with MTX. Only if the patient does not respond to MTX is an anti-TNF drug used. Anti-TNF drugs often result in profound disease improvement, but unfortunately, they can have toxic side effects and are expensive.

For people whose poly JIA is inactive or minimally active on MTX or anti-TNF drugs, 50% to 80% experience a worsening of symptoms once they stop taking the medications. Most of these flare-ups occur within 8 months of stopping treatment. Currently, there is no way to predict which people with poly JIA can safely stop anti-TNF medications. This study will evaluate two different factors-levels of certain calcium binding proteins and production of TNF-for their use in predicting whether people with poly JIA are likely to experience a disease flare-up once they stop anti-TNF treatment. The study will also look for genetic markers that can serve as predictors of safe discontinuation of anti-TNF treatment.

Participation in this study will last up to 14 months and involve up to nine study visits. Visits will be conducted at study entry and after 3, 6, 7, 8, 9, 10, 12, and 14 months. The first three study visits will involve tests to determine baseline health indicators and to ensure inactive disease. If, after 6 months, participants continue to have inactive disease, they will be taken off their anti-TNF medications. For the remainder of the study, visits will be used to monitor disease activity. If participants experience any clinically defined disease flare-ups, they will immediately stop participating in the study and begin additional treatment as prescribed by their health care providers. At all study visits, participants will undergo a general physical examination, a joint examination, questionnaires about how the disease affects their lives, and blood collection for research samples.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of polyarticular JIA (rheumatoid factor + and rheumatoid factor -) or extended oligo JIA by the International League of Associations for Rheumatology (ILAR) criteria
* Receiving therapy with one of the currently available anti-TNF biologics: infliximab, etanercept, or adalimumab
* Absence of any of the FDA label exclusions for anti-TNF therapy
* Receiving slit lamp exams performed at regular intervals in accordance with the published American Academy of Pediatrics guidelines
* Baseline hemoglobin >10 g/dl
* Absence of joints with active arthritis, using the American College of Rheumatology (ACR) definition of "active joint"
* Absence of fever, rash, serositis, splenomegaly, or generalized lymphadenopathy attributable to JIA
* Absence of active uveitis, as per an exam by an ophthalmologist
* Normal erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP); if above normal range, must be not attributable to JIA
* Physician's global assessment of disease activity indicating absence of disease activity, defined as the best score obtainable on the scale used
* Duration of morning stiffness less than or equal to 15 minutes

Exclusion Criteria:

* Diagnosis of a type of JIA other than polyarticular JIA
* Diagnosis of another inflammatory disease that may affect laboratory results or ability to discontinue anti-TNF biologic therapy
* Concurrent treatment with any biologic agent other than infliximab, etanercept, or adalimumab
* previous treatment with rituximab
* concurrent treatment for JIA with corticosteroids >0.2 mg/kg/day OR >10 mg/day

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2009-06; Primary Completion 2013-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Disease flare, defined as demonstrating at least a 30% worsening in at least 3 of the 6 JIA Core Set parameters with no more than 1 improving by more than 30% | Measured at nine study visits over 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Lovell, MD, Principal Investigator — CCHMC
Locations (16):
- United States (16):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Comer Children's Hospital University of Chicago, Chicago, Illinois
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Joseph M Sanzari Children's Hospital, Hackensack, New Jersey
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
deidentified subject information and results of testing have already been shared with multiple investigators requesting samples

REFERENCES:
- [Derived] Hinze CH, Foell D, Johnson AL, Spalding SJ, Gottlieb BS, Morris PW, Kimura Y, Onel K, Li SC, Grom AA, Taylor J, Brunner HI, Huggins JL, Nocton JJ, Haines KA, Edelheit BS, Shishov M, Jung LK, Williams CB, Tesher MS, Costanzo DM, Zemel LS, Dare JA, Passo MH, Ede KC, Olson JC, Cassidy EA, Griffin TA, Wagner-Weiner L, Weiss JE, Vogler LB, Rouster-Stevens KA, Beukelman T, Cron RQ, Kietz D, Schikler K, Mehta J, Ting TV, Verbsky JW, Eberhard AB, Huang B, Giannini EH, Lovell DJ. Serum S100A8/A9 and S100A12 Levels in Children With Polyarticular Forms of Juvenile Idiopathic Arthritis: Relationship to Maintenance of Clinically Inactive Disease During Anti-Tumor Necrosis Factor Therapy and Occurrence of Disease Flare After Discontinuation of Therapy. Arthritis Rheumatol. 2019 Mar;71(3):451-459. doi: 10.1002/art.40727. Epub 2019 Jan 24. PMID 30225949
- [Derived] Lovell DJ, Johnson AL, Huang B, Gottlieb BS, Morris PW, Kimura Y, Onel K, Li SC, Grom AA, Taylor J, Brunner HI, Huggins JL, Nocton JJ, Haines KA, Edelheit BS, Shishov M, Jung LK, Williams CB, Tesher MS, Costanzo DM, Zemel LS, Dare JA, Passo MH, Ede KC, Olson JC, Cassidy EA, Griffin TA, Wagner-Weiner L, Weiss JE, Vogler LB, Rouster-Stevens KA, Beukelman T, Cron RQ, Kietz D, Schikler K, Schmidt KM, Mehta J, Wahezi DM, Ting TV, Verbsky JW, Eberhard BA, Spalding S, Chen C, Giannini EH. Risk, Timing, and Predictors of Disease Flare After Discontinuation of Anti-Tumor Necrosis Factor Therapy in Children With Polyarticular Forms of Juvenile Idiopathic Arthritis With Clinically Inactive Disease. Arthritis Rheumatol. 2018 Sep;70(9):1508-1518. doi: 10.1002/art.40509. Epub 2018 Jul 25. PMID 29604189